CLINICAL TRIAL: NCT05631639
Title: Detection of Upper Gastrointestinal (GI) Bleeding Using a Novel Bleeding Sensor Capsule -A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EnteraSense Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIP-019-01
Record Dates: First submitted 2022-11-14; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Upper Gastrointestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PillSense System (Experimental): The device is composed of an orally ingested sensor capsule and a wireless handheld receiver for real-time display of sensor data. The capsule contains a measuring slot for blood entry. The sensor capsule is used for diagnosis in patients with suspected acute bleeding in the upper gastrointestinal tract.
  Interventions: Device: PillSense System

INTERVENTIONS:
Device: PillSense System — The PillSense capsule is a diagnostic capsule equipped with a sensor for in vivo detection of liquid blood and a paired PillSense receiver for result display.

SUMMARY:
This is a multi-center, prospective, non-randomized, open-label, exploratory clinical investigation performed to evaluate safety and effectiveness of the PillSense System when used for detection of blood in the stomach of patients suspected to have an Upper Gastrointestinal Bleed (UGIB).

DETAILED DESCRIPTION:
The PillSense System consists of the PillSense Capsule, an atraumatic, ingestible, and disposable capsule and PillSense Receiver, an external real-time monitor for results display. The PillSense Capsule is a non-invasive, single use device designed to detect blood in the stomach and wirelessly transmit the data to the external PillSense Receiver. The receiver is a handheld device which displays real-time information gathered from the capsule and clearly displays results, "Blood Detected" or "No Blood Detected".

All enrolled participants were admitted for suspected UGIB and were required to ingest a PillSense Capsule followed by esophagogastroduodenoscopy (EGD) within 1 hour of PillSense Capsule administration. All Patients underwent standard endoscopy following PillSense Capsule evaluation and results were compared with the PillSense System result, i.e., "Blood Detected" or "No Blood Detected".

The study was also designed to confirm transit of the PillSense Capsule through the GI tract and patient tolerability of the PillSense Capsule.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 -80 years
* Ability to give written informed consent
* Clinical suspicion of bleeding

Exclusion Criteria:

1. Circulatory or hemodynamic instability with a clear need for urgent endoscopy or surgery (systolic blood pressure <100 mmHg,heart rate > 100 / min)
2. Known current stenosis of the GI tract
3. Subject is using a pacemaker or other implantable electrical device
4. Dysphagia or difficulties in swallowing pills the size of the capsule
5. History of achalasia or known esophageal dysmotility
6. History of gastroparesis
7. History of severe constipation (1 bowel movement per week or less)
8. Patients who are currently pregnant or breastfeeding, or intend to become pregnant during the investigation
9. Presence of psychological issues preventing participation
10. Stomach bezoar
11. History of Crohn disease
12. History of diverticulitis
13. History of bowel obstruction
14. Suspected gastrointestinal tumor disease
15. Planned MRI investigation (MRI needed before the capsule is excreted)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Device feasibility | within 30 minutes
  Ability of PillSense Capsule to detect the presence or absence of blood and send the results to the PillSense receiver

SECONDARY OUTCOMES:
Device sensitivity | within 2 hours
  Subjects with positive findings for blood based on PillSense and EGD
Device Specificity | within 2 hours
  Subjects with negative findings for blood based on PillSense and EGD
Safety | up to 3 weeks
  Number of patients that developed device-related adverse event (etc. retention, aspiration or bowel obstruction)

CONTACTS AND LOCATIONS:
Locations (3):
- Czechia (3):
  - Fakultní nemocnice Olomouc (FNOL), Olomouc
  - Fakultní nemocnice Ostrava (FNO), Ostrava
  - Institut klinické a experimentální medicíny (IKEM),, Prague